CLINICAL TRIAL: NCT01967329
Title: Canadian North Helicobacter Pylori (CANHelp) Working Group Treatment Trials
Brief Title: CANHelp Working Group Treatment Trials
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Innovates Health Solutions (Other); ArcticNet (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Karen Goodman, Professor, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00007868
Record Dates: First submitted 2013-10-09; First posted 2013-10-22 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Helicobacter Pylori Infection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Standard Triple, treatment naive (Active Comparator): Standard Triple Therapy for H. pylori:
  Oral twice-daily doses of rabeprazole (20 mg), amoxicillin (1 g) and clarithromycin (500 mg)
  One of two treatments randomly assigned to treatment naive participants in Aklavik
  Interventions: Drug: Standard Triple
- Sequential, treatment naive (Active Comparator): Sequential Therapy for H. pylori:
  Oral twice-daily doses of rabeprazole (20 mg) and amoxicillin (1 g) on days 1-5, and on days 6-10, rabeprazole (20 mg), metronidazole (500 mg) and clarithromycin (500 mg)
  One of two treatments randomly assigned to treatment naive participants in Aklavik, Old Crow, Tuktoyaktuk & Fort McPherson
  Interventions: Drug: Sequential
- Quadruple, treatment naive (Active Comparator): Quadruple Thearpy for H. pylori:
  Oral doses of rabeprazole (20 mg) twice daily, metronidazole (500 mg) three times daily, bismuth subsalicylate (Pepto-Bismol) (2 tablets) four times daily and tetracycline (500 mg) four times daily
  One of two treatments randomly assigned to treatment naive participants in Old Crow, Tuktoyaktuk & Fort McPherson
  Interventions: Drug: Quadruple
- Sequential, previous failure(s) (Active Comparator): Sequential Therapy for H. pylori:
  Oral twice-daily doses of rabeprazole (20 mg) and amoxicillin (1 g) on days 1-5, and on days 6-10, rabeprazole (20 mg), metronidazole (500 mg) and clarithromycin (500 mg)
  One of two treatments randomly assigned to participants who previously failed one or more treatments in Aklavik, Old Crow, Tuktoyaktuk & Fort McPherson
  Interventions: Drug: Sequential
- Quadruple, previous failure(s) (Active Comparator): Quadruple Therapy for H. pylori:
  Oral doses of rabeprazole (20 mg) twice daily, metronidazole (500 mg) three times daily, bismuth subsalicylate (Pepto-Bismol) (2 tablets) four times daily and tetracycline (500 mg) four times daily
  One of two treatments randomly assigned to participants who previously failed treatment in Aklavik, Old Crow, Tuktoyaktuk & Fort McPherson
  Interventions: Drug: Quadruple
- Sequential, clarithromycin-resistant (Active Comparator): Sequential Therapy for H. pylori:
  Oral twice-daily doses of rabeprazole (20 mg) and amoxicillin (1 g) on days 1-5, and on days 6-10, rabeprazole (20 mg), metronidazole (500 mg) and clarithromycin (500 mg)
  One of two treatments randomly assigned to participants with known clarithromycin resistance in Aklavik
  Interventions: Drug: Sequential
- Quadruple, clarithromycin-resistant (Active Comparator): Quadruple Therapy for H. pylori:
  Oral doses of rabeprazole (20 mg) twice daily, metronidazole (500 mg) three times daily, bismuth subsalicylate (Pepto-Bismol) (2 tablets) four times daily and tetracycline (500 mg) four times daily
  One of two treatments randomly assigned to participants with known clarithromycin resistance in Aklavik
  Interventions: Drug: Quadruple

INTERVENTIONS:
Drug: Standard Triple — Oral twice-daily doses of rabeprazole (20 mg), amoxicillin (1 g) and clarithromycin (500 mg)
  Other Names: Standard Triple Therapy for H. pylori; Hp-PAC
  Arms: Standard Triple, treatment naive
Drug: Sequential — Oral twice-daily doses of rabeprazole (20 mg) and amoxicillin (1 g) on days 1-5, and on days 6-10, rabeprazole (20 mg), metronidazole (500 mg) and clarithromycin (500 mg)
  Other Names: Sequential Therapy for H. pylori
  Arms: Sequential, clarithromycin-resistant; Sequential, previous failure(s); Sequential, treatment naive
Drug: Quadruple — Oral doses of rabeprazole (20 mg) twice daily, metronidazole (500 mg) three times daily, bismuth subsalicylate (Pepto-Bismol) (2 tablets) four times daily and tetracycline (500 mg) four times daily
  Other Names: Quadruple Therapy for H. pylori
  Arms: Quadruple, clarithromycin-resistant; Quadruple, previous failure(s); Quadruple, treatment naive

SUMMARY:
The CANHelp Working Group Treatment Trials are part of a comprehensive research program carried out by the Canadian North Helicobacter pylori (CANHelp) Working Group. The treatment component involves a series of community-specific trials designed with community input and varying on the specific treatment regimens and number of treatment arms among other study details.

DETAILED DESCRIPTION:
The CANHelp Working Group is a collaborative team that links University of Alberta researchers with Canadian northern community leaders and health officials in a collaborative effort to investigate H. pylori infection with the goal of finding solutions to community concerns about health risks. The research program uses a community-driven research approach in northern communities to characterize the burden of disease from H. pylori infection and exchange knowledge with community members and decision makers to identify ways to reduce health risks from this infection.

For the participating communities, the treatment trials aim to:

1. Estimate the effectiveness of alternate H. pylori treatment regimens to identify optimal regimens for the local setting
2. Identify factors external to the treatment regimen that influence short- and long-term treatment success

ELIGIBILITY:
Inclusion Criteria:

* Over 15 years of age
* Identified as H. pylori infected with a positive urea breath test and/or biopsy-based evidence of H. pylori infection

Exclusion Criteria:

* Allergy to amoxicillin, metronidazole or clarithromycin
* Antibiotic therapy within 4 weeks prior to randomization
* Pregnant or breastfeeding
* Severe cardio-respiratory, pulmonary, endocrine, hepatic or renal disease

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2008-11; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Post-treatment H. pylori status by urea breath test | A minimum of 10 weeks after participant has completed treatment
  Treatment effectiveness, defined as the probability (average risk) of elimination of H. pylori infection following treatment, measured as the proportion of trial participants with a negative post-treatment urea breath test at least 10 weeks following completion of treatment. Using an intention-to-treat analysis, the denominator for this proportion is the number of trial participants assigned treatment. Using a per-protocol analysis, the denominator for this proportion is the number of trial participants who completed treatment and were tested post-treatment.
  Participants are administered a urea breath test using 13C-labeled urea dissolved in a citric acid solution. We use the following test value classifications for determining the outcome:
  >=4.0 (Positive for H. pylori infection) Between 2.5 and 4.0 (Borderline; repeat test) Between 2.4 and -1.99 (Negative for H. pylori infection) Less than -2.0 (Uncertain test result, repeat test)

SECONDARY OUTCOMES:
Adherence to treatment regimen | An expected average of 1 week after treatment is completed
  Participants are asked to return blister packs with unused medication so skipped doses can be counted. Participants are also interviewed to obtain details about their adherence to the regimen.

OTHER OUTCOMES:
Frequency of adverse effects | From the time treatment is started to an expected average of 1 week after treatment is completed
  Participants are contacted by telephone during the completion of the treatment regimen and asked if they have experienced adverse effects. Participants are also interviewed immediately after the completion of treatment and asked if they experienced adverse effects during the completion of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Goodman, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
No plan to make individual participant data (IPD) available

REFERENCES:
- See also: Canadian North Helicobacter pylori (CANHelp) Working Group website — http://www.canhelpworkinggroup.ca/